CLINICAL TRIAL: NCT06319989
Title: The Efficacy of Biplane Versus Single Plane Ultrasound in Facilitating Caudal Epidural Anesthesia in Pediatric Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202301905
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Educational Problems
Keywords: biplane ultrasound; Caudal epidural anesthesia; single plane ultrasound

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel study to assess the efficacy of biplane ultrasound-guided caudal epidural anesthesia in pediatric patients.
Masking Description: The intervention group will receive caudal epidural block under the guidance of biplane ultrasound. The procedures for patients in the control group will be guided by conventional single-plane ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biplane Ultrasound (Other): The intervention group will receive caudal epidural block under the guidance of biplane ultrasound.
  Interventions: Other: Biplane Ultrasound
- Single plane Ultrasound (Other): The procedures for patients in the control group will be guided by conventional single-plane ultrasound.
  Interventions: Other: Single plane ultrasound

INTERVENTIONS:
Other: Biplane Ultrasound — During a standard of care caudal epidural block, biplane ultrasound will be used.
  Arms: Biplane Ultrasound
Other: Single plane ultrasound — During a standard of care caudal epidural block, single plane ultrasound will be used.
  Arms: Single plane Ultrasound

SUMMARY:
Ultrasound guidance plays a pivotal role in caudal epidural block in pediatric patients. In comparison to conventional single-plane ultrasound, biplane ultrasound offers the advantage of providing simultaneous transverse and longitudinal imaging. Better visualization under biplane ultrasound is postulated to enhance the efficacy of caudal epidural blocks. This improvement is expected to manifest through higher first puncture success rate, shorter procedure time, and longer time to first postoperative analgesics use.

DETAILED DESCRIPTION:
Our study aims to recruit pediatric patients receiving caudal epidural blocks as a complement to general anesthesia and for postoperative analgesia. Through a randomized allocation, we will administer the caudal injection with either a biplane ultrasound-guided approach or the single-plane ultrasound-guided technique. The assessment will encompass accuracy metrics, such as the first puncture success rate and number of needle redirections, and the efficiency indicators, including the time from initial probe placement on the skin to successful injection, the time to first postoperative analgesics use, and PACU pain score. Safety evaluation will be conducted, encompassing adverse events from the commencement of the caudal block procedure until discharge. We will also conduct post-discharge follow-up phone calls to evaluate patients' experience after discharge.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II
* Male patients aged 4 months to 10 years
* To undergo elective circumcision with caudal epidural anesthesia as an adjuvant to general anesthesia and for postoperative analgesia

Exclusion Criteria:

* Anatomical anomalies (e.g., tethered cord, sacral malformations, etc.).
* Potential coagulopathy.
* Preoperative analgesics use.
* Allergy to local anesthetics.
* Rash or infection at the injection site.
* Female patients
* Parents refuse to participate.

Ages: 4 Months to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Only male patients would be undergoing elective circumcision with caudal epidural anesthesia as an adjuvant to general anesthesia and for postoperative analgesia.
Enrollment: 281 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
First puncture success | 1 day
  The epidural is obtained on first attempt.

SECONDARY OUTCOMES:
Number of Needle redirections | 1day
  Redirection was defined as pulling the needle back and changing the direction without exiting the skin.
Duration of epidural | 1 day
  Duration from placing the US probe on skin to successful injection (continuous outcome, measured in second).
Postoperative analgesic use | 24 hours post-op
  The time from arriving at PACU to first postoperative analgesics use within 24 hours after discharge (continuous outcome, measured in hour).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Mehta, MS, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States